CLINICAL TRIAL: NCT00279045
Title: A Randomized, Double-Blind Study to Compare the Durability of Glucose Lowering and Preservation of Pancreatic Beta-Cell Function of Rosiglitazone Monotherapy Compared to Metformin or Glyburide/Glibenclamide in Patients With Drug-Naive, Recently Diagnosed Type 2 Diabetes Mellitus
Brief Title: Diabetes Study With Rosiglitazone Monotherapy Versus Metformin Or Glyburide/Glibenclamide
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 49653/048
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: type 2 diabetes monotherapy treatment naive
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Rosiglitazone; Glyburide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Rosiglitazone
Drug: glyburide
Drug: metformin
  Other Names: glyburide; Rosiglitazone

SUMMARY:
The study will compare and evaluate the effects of long-term treatment of monotherapy with rosiglitazone, metformin and glyburide/glibenclamide on the improvement and maintenance of glycemic control in patients with recently diagnosed type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion criteria:

* Newly diagnosed patients (< 3years) with type 2 diabetes.
* Fasting plasma glucose (FPG) range of 126-240 mg/dL at Screening.
* No previous treatment with oral or parenteral glucose-lowering therapy.

Exclusion criteria:

* History of lactic acidosis.
* Anemia (<11g for males, <10 g for females).
* Unstable or severe NY Heart Association-class 3 or 4.
* Any NY Heart Association congestive heart failure.
* Patients with chronic diseases requiring periodic or intermittent treatment with oral or intravenous corticosteroids.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4426 (Actual)
Dates: Start 2000-01-03; Primary Completion 2006-06-01 (Actual); Study Completion 2006-06-19 (Actual)

PRIMARY OUTCOMES:
Time from randomization to the primary action point (monotherapy failure).

SECONDARY OUTCOMES:
Comparison of effects of long-term treatment with Rosiglitazone, Metformin, Glyburide: - maintenance/restoration of beta-cell function: HOMA IS, progression of microalbuminuria, fibrinolytic markers (PAI-1,fibrinogen, CRP).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (418):
- United States (135):
  - GSK Investigational Site, Anniston, Alabama
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Berkeley, California
  - GSK Investigational Site, Corona, California
  - GSK Investigational Site, Fair Oaks, California
  - GSK Investigational Site, Fremont, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Fullerton, California
  - GSK Investigational Site, Greenbrae, California
  - GSK Investigational Site, Harbor City, California
  - GSK Investigational Site, Healdsburg, California
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Loma Linda, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Modesto, California
  - GSK Investigational Site, Pasadena, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Santa Rosa, California
  - GSK Investigational Site, Sunnyvale, California
  - GSK Investigational Site, Ukiah, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Yorba Linda, California
  - GSK Investigational Site, Boulder, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Englewood, Colorado
  - GSK Investigational Site, Longmont, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Palm Harbor, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Titusville, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Blue Ridge, Georgia
  - GSK Investigational Site, Dunwoody, Georgia
  - GSK Investigational Site, Fayetteville, Georgia
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Gurnee, Illinois
  - GSK Investigational Site, Springfield, Illinois
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Lake Charles, Louisiana
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Slidell, Louisiana
  - GSK Investigational Site, Bangor, Maine
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Lansing, Michigan
  - GSK Investigational Site, Royal Oak, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Olive Branch, Mississippi
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Billings, Montana
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Cherry Hill, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Endwell, New York
  - GSK Investigational Site, Flushing, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Mogadore, Ohio
  - GSK Investigational Site, Westlake, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Bend, Oregon
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Downingtown, Pennsylvania
  - GSK Investigational Site, Feasterville, Pennsylvania
  - GSK Investigational Site, Fleetwood, Pennsylvania
  - GSK Investigational Site, Hermitage, Pennsylvania
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, Jefferson Hills, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Upland, Pennsylvania
  - GSK Investigational Site, Warminster, Pennsylvania
  - GSK Investigational Site, West Chester, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Beaumont, Texas
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Irving, Texas
  - GSK Investigational Site, Midland, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Ogden, Utah
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Newport News, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Salem, Virginia
  - GSK Investigational Site, Federal Way, Washington
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Wenatchee, Washington
  - GSK Investigational Site, Charleston, West Virginia
  - GSK Investigational Site, Huntington, West Virginia
  - GSK Investigational Site, Madison, Wisconsin
  - GSK Investigational Site, Milwaukee, Wisconsin
  - GSK Investigational Site, Oregon, Wisconsin
- Austria (2):
  - GSK Investigational Site, Vienna
  - GSK Investigational Site, Wiener Neustadt
- Belgium (9):
  - GSK Investigational Site, Blankenberge
  - GSK Investigational Site, Boechout
  - GSK Investigational Site, Deurne
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Lubbeek (Linden)
  - GSK Investigational Site, Tielt
  - GSK Investigational Site, Wezembeek-Oppem
  - GSK Investigational Site, Wijnegem
  - GSK Investigational Site, Zemst
- Canada (36):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Red Deer, Alberta
  - GSK Investigational Site, Coquitlam, British Columbia
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Victoria, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Cambellton, New Brunswick
  - GSK Investigational Site, Moncton, New Brunswick
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Antigonish, Nova Scotia
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Burlington, Ontario
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Kingston, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Oakville, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Thornhill, Ontario
  - GSK Investigational Site, Thunder Bay, Ontario
  - GSK Investigational Site, Timmins, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Windsor, Ontario
  - GSK Investigational Site, Charlottetown, Prince Edward Island
  - GSK Investigational Site, Chicoutimi, Quebec
  - GSK Investigational Site, La Malbaie, Quebec
  - GSK Investigational Site, Laval, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Plessisville, Quebec
  - GSK Investigational Site, Saint-Marc-des-Carrieres, Quebec
  - GSK Investigational Site, Sainte-Foy, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, St-Isidore de Dorchester, Quebec
  - GSK Investigational Site, Regina, Saskatchewan
  - GSK Investigational Site, Saskatoon, Saskatchewan
- Czechia (5):
  - GSK Investigational Site, Ostrava
  - GSK Investigational Site, Phaha 5
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Ústí nad Labem
  - GSK Investigational Site, Zlín
- Denmark (2):
  - GSK Investigational Site, Frederiksberg C
  - GSK Investigational Site, Odense
- Finland (5):
  - GSK Investigational Site, Hanko
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jyväskylä
  - GSK Investigational Site, Lmatra
  - GSK Investigational Site, Savitaipale
- France (37):
  - GSK Investigational Site, Alben
  - GSK Investigational Site, Bezier
  - GSK Investigational Site, Bourges
  - GSK Investigational Site, Brogile
  - GSK Investigational Site, Chartres
  - GSK Investigational Site, Denguin
  - GSK Investigational Site, Évreux
  - GSK Investigational Site, Gamarde-les-Bains
  - GSK Investigational Site, La Rochelle
  - GSK Investigational Site, Labarthe-sur-Lèze
  - GSK Investigational Site, Le Mans
  - GSK Investigational Site, Le Pian-Médoc
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Mallemort
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Marsillargues
  - GSK Investigational Site, Marssac-sur-Tarn
  - GSK Investigational Site, Mont de Marsen
  - GSK Investigational Site, Montignac
  - GSK Investigational Site, Moulon
  - GSK Investigational Site, Mûrs-Erigné
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Nîmes
  - GSK Investigational Site, Orthez
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Roanna
  - GSK Investigational Site, Saint Genies Des Fontaines
  - GSK Investigational Site, Saint-Etienne
  - GSK Investigational Site, Saint-Julien-des-Landes
  - GSK Investigational Site, Saint-Martin-d'Hères
  - GSK Investigational Site, Saint-Pierre-de-Chandieu
  - GSK Investigational Site, Sisteron
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Tarare
  - GSK Investigational Site, Vieux-Condé
  - GSK Investigational Site, Vourey
- Germany (59):
  - GSK Investigational Site, Bad Rappenau, Baden-Wurttemberg
  - GSK Investigational Site, Deggingen, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Trochtelfingen, Baden-Wurttemberg
  - GSK Investigational Site, Unterschneidheim, Baden-Wurttemberg
  - GSK Investigational Site, Wangen, Baden-Wurttemberg
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Aschaffenburg, Bavaria
  - GSK Investigational Site, Haag, Bavaria
  - GSK Investigational Site, Höhenkirchen-Siegertsbrunn, Bavaria
  - GSK Investigational Site, Ismaning, Bavaria
  - GSK Investigational Site, Krummenaab, Bavaria
  - GSK Investigational Site, Künzing, Bavaria
  - GSK Investigational Site, Landshut, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Wallerfing, Bavaria
  - GSK Investigational Site, Bad Kreuznach, Hesse
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Großalmerode, Hesse
  - GSK Investigational Site, Lollar, Hesse
  - GSK Investigational Site, Offenbach, Hesse
  - GSK Investigational Site, Schaafheim, Hesse
  - GSK Investigational Site, Vellmar, Hesse
  - GSK Investigational Site, Damme, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Hildesheim, Lower Saxony
  - GSK Investigational Site, Lüneburg, Lower Saxony
  - GSK Investigational Site, Paderborn, Lower Saxony
  - GSK Investigational Site, Winsen/Lohe, Lower Saxony
  - GSK Investigational Site, Beckum, North Rhine-Westphalia
  - GSK Investigational Site, Bergkamen, North Rhine-Westphalia
  - GSK Investigational Site, Borken, North Rhine-Westphalia
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Duisburg, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Euskirchen, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Lüdenscheid, North Rhine-Westphalia
  - GSK Investigational Site, Lünen, North Rhine-Westphalia
  - GSK Investigational Site, Neuss, North Rhine-Westphalia
  - GSK Investigational Site, Schwabenheim, North Rhine-Westphalia
  - GSK Investigational Site, Siegen, North Rhine-Westphalia
  - GSK Investigational Site, Warendorf, North Rhine-Westphalia
  - GSK Investigational Site, Deidesheim, Rhineland-Palatinate
  - GSK Investigational Site, Diez, Rhineland-Palatinate
  - GSK Investigational Site, Lambrecht, Rhineland-Palatinate
  - GSK Investigational Site, Rhaunen, Rhineland-Palatinate
  - GSK Investigational Site, Chemnitz, Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Freital, Saxony
  - GSK Investigational Site, Pirna, Saxony
  - GSK Investigational Site, Schmiedeberg, Saxony
  - GSK Investigational Site, Itzehoe, Schleswig-Holstein
  - GSK Investigational Site, Ratzeburg, Schleswig-Holstein
  - GSK Investigational Site, Wahlstedt, Schleswig-Holstein
  - GSK Investigational Site, Wilster, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Hungary (2):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Miskolc
- Ireland (6):
  - GSK Investigational Site, Belfast
  - GSK Investigational Site, Co. Tipperary
  - GSK Investigational Site, Cork
  - GSK Investigational Site, Dublin
  - GSK Investigational Site, Gowran
  - GSK Investigational Site, Kilkenny
- Italy (22):
  - GSK Investigational Site, Acquaviva Delle Fonti (BA), Apulia
  - GSK Investigational Site, Ferrara, Emilia-Romagna
  - GSK Investigational Site, Ravenna, Emilia-Romagna
  - GSK Investigational Site, Scandiano (RE), Emilia-Romagna
  - GSK Investigational Site, Rozzano (MI), Lombardy
  - GSK Investigational Site, Catania, Sicily
  - GSK Investigational Site, Città Di Castello (PG), Umbria
  - GSK Investigational Site, Florence
  - GSK Investigational Site, La Spezia
  - GSK Investigational Site, Lecce
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Palermo
  - GSK Investigational Site, Parma
  - GSK Investigational Site, Perugia
  - GSK Investigational Site, Rovigo
  - GSK Investigational Site, S. Benedetto TR (AP)
  - GSK Investigational Site, San Giovanni Rotondo FG
  - GSK Investigational Site, Sassari
  - GSK Investigational Site, Terni
  - GSK Investigational Site, Torino
  - GSK Investigational Site, Udine
  - GSK Investigational Site, Vicenza
- Netherlands (9):
  - GSK Investigational Site, 's-Hertogenbosch
  - GSK Investigational Site, De Bilt
  - GSK Investigational Site, Geleen
  - GSK Investigational Site, Hengelo
  - GSK Investigational Site, Huizen
  - GSK Investigational Site, Losser
  - GSK Investigational Site, Rijswijk
  - GSK Investigational Site, Roelofarendsveen
  - GSK Investigational Site, Woerden
- Norway (3):
  - GSK Investigational Site, Hamar
  - GSK Investigational Site, Paradis
  - GSK Investigational Site, Skedsmokorset
- Spain (37):
  - GSK Investigational Site, Albaida (Valencia)
  - GSK Investigational Site, Basurto/Bilbao
  - GSK Investigational Site, Benassal (Castellón)
  - GSK Investigational Site, Benicasim (Castellón)
  - GSK Investigational Site, Bilbao
  - GSK Investigational Site, Cartagena
  - GSK Investigational Site, Cáceres
  - GSK Investigational Site, El Palmar (Murcia)
  - GSK Investigational Site, Elche (Alicante)
  - GSK Investigational Site, Elda-Alicante
  - GSK Investigational Site, Figueras
  - GSK Investigational Site, Girona
  - GSK Investigational Site, Granollers (Barcelona)
  - GSK Investigational Site, Jerez (Cadiz)
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Mataró
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Mérida
  - GSK Investigational Site, Olleria, Valencia
  - GSK Investigational Site, Onda/Castellón
  - GSK Investigational Site, Orihuela (Alicante)
  - GSK Investigational Site, Plasencia
  - GSK Investigational Site, Pontevedra
  - GSK Investigational Site, Sagunto/Valencia
  - GSK Investigational Site, San Juan (Alicante)
  - GSK Investigational Site, San Vincente Raspeig (Alicante)
  - GSK Investigational Site, Santa Coloma de Gramanet (Barcelona)
  - GSK Investigational Site, Santa Cruz de Tenerife
  - GSK Investigational Site, Tereul
  - GSK Investigational Site, Toledo
  - GSK Investigational Site, Torrelavega/Santander
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Valladolid
  - GSK Investigational Site, Vallda (Valencia)
  - GSK Investigational Site, Villajoyosa - Alicante
  - GSK Investigational Site, Zamora
  - GSK Investigational Site, Zaragoza
- Sweden (5):
  - GSK Investigational Site, Älta
  - GSK Investigational Site, Degerberga
  - GSK Investigational Site, Gimo
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Stockholm
- United Kingdom (44):
  - GSK Investigational Site, Aberdeen, Aberdeenshire
  - GSK Investigational Site, Sandy, Bedfordshire
  - GSK Investigational Site, Reading, Berkshire
  - GSK Investigational Site, Llanelli, Carmarthenshire
  - GSK Investigational Site, Warrington, Cheshire
  - GSK Investigational Site, Bournemouth, Dorset
  - GSK Investigational Site, Poole, Dorset
  - GSK Investigational Site, Barry, Glamorgan
  - GSK Investigational Site, Cardiff, Glamorgan
  - GSK Investigational Site, Hemel Hempstead, Hertfordshire
  - GSK Investigational Site, Stevenage, Hertfordshire
  - GSK Investigational Site, Airdrie, Lanarkshire
  - GSK Investigational Site, Glasgow, Lanarkshire
  - GSK Investigational Site, Bolton, Lancashire
  - GSK Investigational Site, Chorley, Lancashire
  - GSK Investigational Site, Edinburgh, Midlothian
  - GSK Investigational Site, Wellingborough, Northamptonshire
  - GSK Investigational Site, Nottingham, Nottinghamshire
  - GSK Investigational Site, Haverfordwest, Pembrokeshire
  - GSK Investigational Site, Frome, Somerset
  - GSK Investigational Site, Crawley, Sussex West
  - GSK Investigational Site, Nuneaton, Warwickshire
  - GSK Investigational Site, Rugby, Warwickshire
  - GSK Investigational Site, Livingston, West Lothian
  - GSK Investigational Site, Melksham, Wiltshire
  - GSK Investigational Site, Trowbridge, Wiltshire
  - GSK Investigational Site, Barnsley
  - GSK Investigational Site, Bath
  - GSK Investigational Site, Bradford
  - GSK Investigational Site, Cardiff
  - GSK Investigational Site, Co.Antrim
  - GSK Investigational Site, Doncaster
  - GSK Investigational Site, Gateshead
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Glenrothes
  - GSK Investigational Site, Irvine
  - GSK Investigational Site, Kent
  - GSK Investigational Site, Leicester
  - GSK Investigational Site, London
  - GSK Investigational Site, Newtownabbey
  - GSK Investigational Site, Peterborough
  - GSK Investigational Site, Swansea
  - GSK Investigational Site, Wakefield
  - GSK Investigational Site, Wigan

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Viberti G, Kahn SE, Greene DA, Herman WH, Zinman B, Holman RR, Haffner SM, Levy D, Lachin JM, Berry RA, Heise MA, Jones NP, Freed MI. A diabetes outcome progression trial (ADOPT): an international multicenter study of the comparative efficacy of rosiglitazone, glyburide, and metformin in recently diagnosed type 2 diabetes. Diabetes Care. 2002 Oct;25(10):1737-43. doi: 10.2337/diacare.25.10.1737. PMID 12351470
- [Result] Viberti G, Lachin J, Holman R, Zinman B, Haffner S, Kravitz B, Heise MA, Jones NP, O'Neill MC, Freed MI, Kahn SE, Herman WH; ADOPT Study Group. A Diabetes Outcome Progression Trial (ADOPT): baseline characteristics of Type 2 diabetic patients in North America and Europe. Diabet Med. 2006 Dec;23(12):1289-94. doi: 10.1111/j.1464-5491.2006.02022.x. PMID 17116177
- [Result] Kahn SE, Haffner SM, Heise MA, Herman WH, Holman RR, Jones NP, Kravitz BG, Lachin JM, O'Neill MC, Zinman B, Viberti G; ADOPT Study Group. Glycemic durability of rosiglitazone, metformin, or glyburide monotherapy. N Engl J Med. 2006 Dec 7;355(23):2427-43. doi: 10.1056/NEJMoa066224. Epub 2006 Dec 4. PMID 17145742
- [Result] Kahn SE, Zinman B, Haffner SM, O'Neill MC, Kravitz BG, Yu D, Freed MI, Herman WH, Holman RR, Jones NP, Lachin JM, Viberti GC; ADOPT Study Group. Obesity is a major determinant of the association of C-reactive protein levels and the metabolic syndrome in type 2 diabetes. Diabetes. 2006 Aug;55(8):2357-64. doi: 10.2337/db06-0116. PMID 16873701
- [Result] Zinman B, Kahn SE, Haffner SM, O'Neill MC, Heise MA, Freed MI; ADOPT Study Group. Phenotypic characteristics of GAD antibody-positive recently diagnosed patients with type 2 diabetes in North America and Europe. Diabetes. 2004 Dec;53(12):3193-200. doi: 10.2337/diabetes.53.12.3193. PMID 15561950
- [Derived] El-Damanawi R, Stanley IK, Staatz C, Pascoe EM, Craig JC, Johnson DW, Mallett AJ, Hawley CM, Milanzi E, Hiemstra TF, Viecelli AK. Metformin for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2024 Jun 4;6(6):CD013414. doi: 10.1002/14651858.CD013414.pub2. PMID 38837240
- [Derived] Gnesin F, Thuesen ACB, Kahler LKA, Madsbad S, Hemmingsen B. Metformin monotherapy for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Jun 5;6(6):CD012906. doi: 10.1002/14651858.CD012906.pub2. PMID 32501595
- [Derived] Lachin JM, Viberti G, Zinman B, Haffner SM, Aftring RP, Paul G, Kravitz BG, Herman WH, Holman RR, Kahn SE; ADOPT Study Group. Renal function in type 2 diabetes with rosiglitazone, metformin, and glyburide monotherapy. Clin J Am Soc Nephrol. 2011 May;6(5):1032-40. doi: 10.2215/CJN.09291010. Epub 2011 Mar 31. PMID 21454723
- [Derived] Kahn SE, Haffner SM, Viberti G, Herman WH, Lachin JM, Kravitz BG, Yu D, Paul G, Holman RR, Zinman B; Diabetes Outcome Progression Trial (ADOPT) Study Group. Rosiglitazone decreases C-reactive protein to a greater extent relative to glyburide and metformin over 4 years despite greater weight gain: observations from a Diabetes Outcome Progression Trial (ADOPT). Diabetes Care. 2010 Jan;33(1):177-83. doi: 10.2337/dc09-1661. Epub 2009 Oct 6. PMID 19808911
- [Derived] Kahn SE, Zinman B, Lachin JM, Haffner SM, Herman WH, Holman RR, Kravitz BG, Yu D, Heise MA, Aftring RP, Viberti G; Diabetes Outcome Progression Trial (ADOPT) Study Group. Rosiglitazone-associated fractures in type 2 diabetes: an Analysis from A Diabetes Outcome Progression Trial (ADOPT). Diabetes Care. 2008 May;31(5):845-51. doi: 10.2337/dc07-2270. Epub 2008 Jan 25. PMID 18223031
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 49653/048 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 49653/048 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 49653/048 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 49653/048 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 49653/048 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 49653/048 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 49653/048 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register